CLINICAL TRIAL: NCT07276893
Title: Preparation of the Pediatric Patient Before Cardiac Catheterization: A Randomized Controlled Trial
Brief Title: Preop Preparation Before Cardiac Catheterization
Acronym: Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/228
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Abnormalities; Preoperative Care; Children; Pediatric Nursing; Animation
Keywords: pediatric nursing; preoperative care; children; animation; cardiac diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: This parallel-group randomized controlled experimental study was designed to determine the effect of showing an animated film using virtual reality glasses to pediatric patients undergoing cardiac catheterization and the routine procedure on surgery-related anxiety, fear, and postoperative pain. Stratified Block Randomization Method were used. 1 (Experimental Group) and 2 (Control Group): The randomizer.org website was used to create the blocks.
Who Masked: Participant
Masking Description: Only participants were masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animated film using virtual reality glasses group (Experimental): Prior to the cardiac catheterization procedure, the researcher administered the Individual Assessment Form and the Children's Fear Scale to the children and had them complete the Children's Anxiety Scale-State Scale. One hour before the procedure, the children were shown the animated film "Super Heart Team: Ready for Action" using virtual reality glasses. After the animated film was shown to the child, the Child Anxiety Scale-State (CAS-D) was administered, and the Child Fear Scale was assessed by the researcher. Thirty minutes after the cardiac catheterization procedure was completed and the child returned to the children's ward, the researcher evaluated the Child Fear Scale and Wong Baker Facial Pain Scale and had the child complete the Child Anxiety Scale-State (CAS-D). Additionally, heart rate, respiratory rate, and O2 saturation were recorded at 15, 30, and 60 min after the procedure.
  Interventions: Behavioral: animated film via virtual reality glasses
- Control group (No Intervention): Prior to cardiac catheterization, the researcher administered the Individual Assessment Form and the Children's Fear Scale to the children and had them complete the Children's Anxiety Scale-State Scale. Children in this group continued to undergo routine procedures at the clinic. Half an hour after the cardiac catheterization procedure was completed and the child returned to the children's ward, the researcher administered the Children's Fear Scale and the Wong Baker Facial Pain Scale and ensured that the child completed the Children's Anxiety Scale, State (CAS-D) Scale. In addition, heart rate, respiratory rate, and O2 saturation were recorded at 15, 30, and 60 min after the procedure.

INTERVENTIONS:
Behavioral: animated film via virtual reality glasses — One hour before the procedure, the children were shown the animated film "Super Heart Team: Ready for Action" using virtual reality glasses.
  Arms: Animated film using virtual reality glasses group

SUMMARY:
This study aimed to determine the effect of an animated film shown through virtual reality (VR) glasses before cardiac catheterization on children's pre-procedure anxiety and fear levels and post-procedure pain. H1: Animated films viewed through virtual reality glasses reduce procedure-related anxiety in children.

H2: Animated films viewed through virtual reality glasses reduce procedure-related fear in children.

H3: Animated films viewed through virtual reality glasses reduce procedure-related pain in children.

Prior to the cardiac catheterization procedure, the researcher administered the Individual Assessment Form and the Children's Fear Scale to the children and had them complete the Children's Anxiety Scale-State Scale. One hour before the procedure, the children were shown the animated film "Super Heart Team: Ready for Action" using virtual reality glasses. After the animated film was shown to the child, the Child Anxiety Scale-State (CAS-D) was administered, and the Child Fear Scale was assessed by the researcher. Thirty minutes after the cardiac catheterization procedure was completed and the child returned to the children's ward, the researcher evaluated the Child Fear Scale and Wong Baker Facial Pain Scale and had the child complete the Child Anxiety Scale-State (CAS-D). Additionally, heart rate, respiratory rate, and O2 saturation were recorded at 15, 30, and 60 min after the procedure.

DETAILED DESCRIPTION:
Healthcare professionals have developed preoperative preparation programs that include methods such as short films, videos, picture books, play activities, and surgical room tours to help children cope with surgical procedures and reduce negative reactions. These methods are low-cost, minimally invasive, have a minimal risk of adverse effects, and are continuously and widely applicable to various diseases. Studies indicate that animated videos used to distract children's attention before surgery reduce preoperative anxiety (Özyılmaz et al., 2024; Yang et al., 2022) and increase compliance during surgery (Yang et al., 2022).

This study aimed to determine the effect of an animated film shown through virtual reality (VR) glasses before cardiac catheterization on children's pre-procedure anxiety and fear levels and post-procedure pain. H1: Animated films viewed through virtual reality glasses reduce procedure-related anxiety in children.

H2: Animated films viewed through virtual reality glasses reduce procedure-related fear in children.

H3: Animated films viewed through virtual reality glasses reduce procedure-related pain in children.

Prior to the cardiac catheterization procedure, the researcher administered the Individual Assessment Form and the Children's Fear Scale to the children and had them complete the Children's Anxiety Scale-State Scale. One hour before the procedure, the children were shown the animated film "Super Heart Team: Ready for Action" using virtual reality glasses. After the animated film was shown to the child, the Child Anxiety Scale-State (CAS-D) was administered, and the Child Fear Scale was assessed by the researcher. Thirty minutes after the cardiac catheterization procedure was completed and the child returned to the children's ward, the researcher evaluated the Child Fear Scale and Wong Baker Facial Pain Scale and had the child complete the Child Anxiety Scale-State.

Control GRoup Prior to cardiac catheterization, the researcher administered the Individual Assessment Form and the Children's Fear Scale to the children and had them complete the Children's Anxiety Scale-State Scale. Children in this group continued to undergo routine procedures at the clinic. Half an hour after the cardiac catheterization procedure was completed and the child returned to the children's ward, the researcher administered the Children's Fear Scale and the Wong Baker Facial Pain Scale and ensured that the child completed the Children's Anxiety Scale, State (CAS-D) Scale. In addition, heart rate, respiratory rate, and O2 saturation were recorded at 15, 30, and 60 min after the procedure.(CAS-D). Additionally, heart rate, respiratory rate, and O2 saturation were recorded at 15, 30, and 60 min after the procedure.

ELIGIBILITY:
Inclusion Criteria

* Being a child patient aged 5-10 years old hospitalized in the Cardiology Clinic of Ege University Hospital (Health Application and Research Center) Children's
* Hospital and scheduled for cardiac catheterization,
* The child being able to read and write,
* Having developed language skills/no communication problems,
* The family agreed to participate in the study,
* The child volunteered to participate in the study, Exclusion Criteria
* Having vision problems or wearing glasses,
* Having a psychological diagnosis,
* Not being able to understand or speak Turkish,
* The child did not want to complete the scales after the procedure,
* The child or parent wanting to withdraw from the study,
* Not agreeing to participate in the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Child Anxiety Scale | One hour before the procedure, 30 minutes after the procedure
  Animated films viewed through virtual reality glasses reduce procedure-related anxiety in children.
Child Fear Scale | one hour before the procedure, 30 minutes after the procedure
  Animated films viewed through virtual reality glasses reduce procedure-related fear in children.
Wong Baker Facial Pain Scale | Thirty minutes after the procedure
  Animated films viewed through virtual reality glasses reduce procedure-related pain in children.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Uzsen, Phd, Principal Investigator — Ondokuz Mayıs University; Dilek Zengin, Phd, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Aegean Sea Zone, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No